CLINICAL TRIAL: NCT00956982
Title: Pegylated Interferon Alpha-2b Plus Ribavirin Combination Treatment for Older Patients With Chronic Hepatitis C
Brief Title: PEG-IFN Plus Ribavirin Combination Therapy for Older Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyushu University (Other)
Responsible Party: Jun Hayashi, Department of General Medicine, Kyushu University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KULDS2009
Record Dates: First submitted 2009-08-06; First posted 2009-08-11 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C Virus Pegylated Interferon Ribavirin Older
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pegylated interferon alpha-2b plus ribavirin — All patients were treated with a weight-based, 1.5 μg/kg weekly dose of subcutaneous PEG-IFN alpha-2b (PegIntron A, Schering-Plough, Osaka, Japan), in combination with PEG-IFN alpha-2b, RBV (Rebetol; Schering-Plough), which was given orally at a daily dose of 600-1000mg based on bodyweight (600 mg for patients weighing < 60 kg, 800 mg for those weighing 60-80 kg, and 1000 mg for those weighing 80 kg). The length of treatment was 48 weeks for patients with HCV of genotype 1and 24 weeks for patients with genotypes 2, respectively

SUMMARY:
The purpose of this study is to analyze the efficacy and safety of a combination therapy of pegylated interferon (PEG-IFN) alpha-2b plus ribavirin (RBV) for older Japanese patients (≧65years old) infected with hepatitis C virus (HCV) compared with younger patients(< 65 years old).

ELIGIBILITY:
Inclusion Criteria:

* A prospective study of 2270 Japanese patients aged 18 years or older treated with PEG-IFN alpha-2b plus RBV was done between December 2004 and July 2008.
* All positive for both antibody to HCV and HCV-RNA for over six months and were enrolled.

Exclusion Criteria:

* Clinical or biochemical evidence of hepatic decompensation.
* Advanced cirrhosis identified by large esophageal varices (F2 or F3).
* History of gastrointestinal bleeding, ascites, encephalopathy, or hepatocellular carcinoma.
* Hemoglobin level < 11.5g/L, white blood cell count < 3×10９/Ｌ，and platelet count < 50×10９/Ｌ.
* Concomitant liver disease other than hepatitis C(hepatitis B surface antigen positive or HIV positive).
* Excessive active alcohol consumption > 60 g/day or drug abuse.
* Severe psychiatric disease.
* Antiviral or corticosteroid therapy within 12 months prior to the enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1251 (Estimated)
Dates: Start 2004-12; Primary Completion 2008-07 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
antiviral effect by PEG-IFN alpha-2b plus RBV treatment | 24-weeks follow-up after the end of treatment

SECONDARY OUTCOMES:
the tolerance of older patients by PEG-IFN alpha-2b plus RBV treatment | during PEG-IFN alpha-2b plus RBV treatment (48 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Hayashi, Principal Investigator — Department of General Medicine, Kyushu University Hospital
Locations (1):
- Department of General Medicine, Kyushu University Hospital, Fukuoka, Japan